CLINICAL TRIAL: NCT07037472
Title: A Cohort Study Establishing a Standardized Scoring System in Dermatomyositis With Calcinosis Cutis and Assessing Treatment Response Via Multimodal Photoacoustic-Ultrasound Imaging
Brief Title: Photoacoustic/Ultrasound Imaging in Patients of Dermatomyositis With Calcinosis Cutis: Characteristic Findings and Treatment Response Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PA/US Dermatomyositis
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-06

CONDITIONS: Dermatomyositis; Dermatomyositis With Calcinosis Cutis
Keywords: Dermatomyositis; Dermatomyositis with Calcinosis cutis; Photoacoustic imaging
MeSH Terms: conditions — Dermatomyositis | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DM with calcinosis disease severity assessment based on PA/US imaging (Experimental): Establish a non-invasive photoacoustic-ultrasound (PA/US) imaging evaluation method for DM with calcinosis to identify the characteristic PA/US manifestations of DM patients with different types of skin lesions, and use PAI to further assess the disease severity of DM patient.
  Interventions: Diagnostic Test: Multi-modal photoacoustic/ultrasonic (PA/US) imaging system
- DM patients with calcinosis planning to undergo drug treatment based on PA/US imaging (Experimental): Patients over 18 years of age with histopathologically or clinically confirmed diagnoses based on the 2017 EULAR/ACR classification criteria who plan to undergo drug treatment.
  Interventions: Drug: Drug treatment

INTERVENTIONS:
Diagnostic Test: Multi-modal photoacoustic/ultrasonic (PA/US) imaging system — The multi-modal PA/US imaging system is equipped with a handheld PA/US probe, and able to provide data of dual-wavelength PA imaging of DM skin lesions, in addition to real-time 2D conventioanl US imaging
  Arms: DM with calcinosis disease severity assessment based on PA/US imaging
Drug: Drug treatment — The multi-modal PA/US imaging system is equipped with a handheld PA/US probe, and able to provide data of dual-wavelength PA imaging of DM skin lesions, in addition to real-time 2D conventional US imaging. The histopathological biopsy results before and after treatment are combined as indicators for evaluating therapeutic efficacy and predicting treatment outcomes.
  Arms: DM patients with calcinosis planning to undergo drug treatment based on PA/US imaging

SUMMARY:
Photoacoustic imaging (PAI) is an emerging biomedical modality that integrates the advantages of optical contrast and ultrasound imaging depth. Capable of providing morphological, functional, and molecular information, PAI shows significant promise for visualizing human superficial tissue. The goal of this clinical trial is to build a PAI evaluation method for DM skin lesions, explore its application value in assessing DM disease severity and evaluation of treatment response. The main questions it aims to answer are:

1. How to establish a non-invasive PA/US imaging evaluation method for DM skin lesions?
2. Can PAI precisely assess DM disease severity?
3. Can PAI systems predict the treatment response in DM with calcinosis cutis? Participants will receive regular PA/US imaging examinations during five stages of treatment (before treatment, 3 months, 6 months, 9 months and 12 months). And the effectiveness of PA/US in treatment response for DM at different time points will be evaluated.

DETAILED DESCRIPTION:
A multimodal photoacoustic-ultrasound (PA/US) system was integrated into a high-end commercial US platform, enabling real-time acquisition of grayscale imaging, color Doppler (CDUS), and dual-wavelength photoacoustic (PAI) data. The PA/US images were acquired using a hand-held probe integrated optical devices and US transducers. Researchers plan to recruit participants of DM with calcinosis cutis from the department of rheumatology in Peking Union Medical College Hospital. The patients are scheduled to receive multi-modality PA/US imaging examinations, which integrated gray scale ultrasound (GSUS), ultra-micro-angiography (UMA) and PAI to realize visualization and assessment of subcutaneous soft tissues in morphology, hemodynamics, blood flow and oxygenation. This clinical trial aims to address three key objectives: the establishment of a non-invasive PA/US imaging evaluation method for DM skin lesions, the applicaiton to assess DM disease severity, and the use of PAI to monitor the treatment response.

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilled the 2017 EULAR/ACR classification criteria for idiopathic inflammatory myositis. Of the adult DM patients enrolled, those were found to have calcinosis and were subsequently included in our analysis.
* Among enrollees with idiopathic inflammatory myositis, patients with pathognomonic skin rashes were subclassified as DM or amyopathic DM patients based on the 2017 EULAR/ACR classification tree.
* For patients without pathognomonic skin manifestations, DM was defined according to muscle biopsy.
* Patients with amyopathic DM were grouped with DM patients.
* Calcinosis diagnosis was based on clinical examination findings.

Exclusion Criteria:

* Patients whose age at disease onset was <18 years and those with overlap syndrome and/or IBM were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify photoacoustic features of skin lesions of DM with calcinosis and establish PA/US Scoring System for assessing disease severity of DM | From enrollment to the end of treatment at 2 year
  Photoacoustic excitation and photoacoustic imaging detection will be performed
Predict the treatment response of DM with calcinosis Using PA/US Parameters | From enrollment to the end of treatment at 2 year
  PA/US Scoring System will be used for assessing changes of DM disease severity after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided